CLINICAL TRIAL: NCT01222650
Title: A Randomized, Double-blind, Placebo-controlled, Multicentre Study of KSO-0400 in BPH Patients With LUTS
Brief Title: A Comparative Study of KSO-0400 in BPH Patients With LUTS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kissei Pharmaceutical Co., Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KSO1201
Record Dates: First submitted 2010-10-15; First posted 2010-10-18 (Estimated); Last update posted 2011-07-04 (Estimated); Status verified 2011-06

CONDITIONS: Benign Prostatic Hyperplasia (BPH)
Keywords: Benign Prostatic Hyperplasia; I-PSS; α1A-AR antagonist
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — silodosin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- KSO-0400 Low Dose (Experimental)
  Interventions: Drug: KSO-0400
- KSO-0400 High Dose (Experimental)
  Interventions: Drug: KSO-0400
- Silodosin (Experimental)
  Interventions: Drug: Silodosin
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: KSO-0400
  Arms: KSO-0400 Low Dose
Drug: KSO-0400
  Arms: KSO-0400 High Dose
Drug: Silodosin
  Arms: Silodosin
Drug: Placebo
  Arms: Placebo

SUMMARY:
The objective of this study is to evaluate the efficacy and safety of KSO-0400 compared to placebo for the treatment of LUTS caused by BPH.

ELIGIBILITY:
Inclusion Criteria:

* BPH patients with LUTS

Exclusion Criteria:

* Patients with a history of prostatectomy, intrapelvic radiation therapy, thermotherapy of prostate or prostatic hyperthermia
* Patients with prostate cancer or suspected prostate cancer
* Patients who have any clinically relevant cardiovascular, hepatic or renal disorder

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400

PRIMARY OUTCOMES:
Change in I-PSS Total Score from baseline | Baseline and 12 weeks (LOCF)

SECONDARY OUTCOMES:
Change in I-PSS Sub-score from baseline | Baseline and 12 weeks (LOCF)
Change in QOL Score from baseline | Baseline and 12 weeks (LOCF)
Change in Qmax (maximum urinary flow rate) from baseline | Baseline and 12 weeks (LOCF)

CONTACTS AND LOCATIONS:
Overall Officials: Katsumi Hontani, Study Director — Clinical Development Dept.,Kissei Pharmaceutical Co., Ltd.
Locations (1):
- Japan, Kanto Region, Japan